CLINICAL TRIAL: NCT05640492
Title: Metacognitive Training in the Older Adults With Depressive Symptoms
Brief Title: Metacognitive Training in the Older Adults With Depressive Symptoms (MCT-Silver)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Évora (Other)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Lara Manuela Guedes de Pinho, Principal Investigator, University of Évora
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GD/29805/2022
Record Dates: First submitted 2022-10-06; First posted 2022-12-07 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Depressive Symptoms
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MCT Group (Experimental): Older adults (more than 59 years old) with depressive symptoms
  Interventions: Behavioral: Metacognitive Training for Depression in Later Life (MCT-Silver)
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Metacognitive Training for Depression in Later Life (MCT-Silver) — MCT-Silver consists of eight modules, each of which begins with psychoeducational and "normalizing" elements. A mastery is presented through examples and exercises, and the fallibility of human cognition is discussed and illustrated. In a second phase, the pathological extremes of each cognitive bias are highlighted and the participant is shown how the exacerbation of (normal) thinking biases can lead to problems in daily life. It is intended with this exercise that participants learn how to identify and mitigate cognitive "traps". Dysfunctional coping strategies (social isolation and negative thoughts) are highlighted, and suggestions for replacing them with adaptive strategies are given. Homework assignments are distributed at the end of each session (Schneider et al., 2018).
  Arms: MCT Group

SUMMARY:
Depression is one of the most common mental disorders in older adults and a major cause of years lived with disability. Depression does not always respond to antidepressants, and non-pharmacological interventions are recommended by international guidelines. The Metacognitive Training for Depression in Later Life (MCT-Silver) is a creative and innovative group intervention that aims to reduce depressive symptoms by challenging the cognitive and metacognitive beliefs characteristic of this disorder, that intends to enable participants to recognize and correct their automatic and dysfunctional thinking patterns and behavior. It was developed by the partner institution's team, and has already demonstrated positive results. This project aims to extend the research study to Portugal, through cultural adaptation, pilot study, and a Randomized Controlled Trial (RCT). To this end, we defined the following aims: To plan and conduct a pilot study to assess the efficacy of the MCT-Silver in the Portuguese population; To conduct a multicenter randomized controlled trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Age: 60 years or older
* Sufficient command of the Portuguese language
* Willingness to participate in the intervention for a period of 4 to 8 weeks (participants who do not participate in the intervention will also be included in the analysis)
* Adequate visual and hearing acuity for neuropsychological testing and participation in the group sessions
* Values above 10 on the Hamilton Depression Scale

Exclusion Criteria:

* Active psychotic symptoms (i.e., hallucinations, delusions, or manias)
* Acute suicidal ideation
* Cognitive impairment
* Dementia or other neurological disease

Ages: 60 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HRSD-24) | Baseline
  The 24-item version of the Hamilton Depression Rating Scale is an established clinician-rated assessment of depressive symptom severity and assesses psychological as well as somatic symptoms (scores range from 0-2 or 0-4) of depression. The clinician rates the severity of these symptoms based on the patient's report and his or her own observation. Scores range from 0-54. Based on the first 17 items, a score of 8-13 indicates mild depression, 14-18 indicates moderate depression, 19-22 indicates severe depression and scores greater than 23 indicate very severe depression. The scale has demonstrated good sensitivity and specificity among older adults (Mottram, Wilson & Copeland, 2001). The reliability and validity among older adult samples has also been confirmed (Korner et al., 2006). In terms of assessing change for the current trial, a greater reduction in depressive symptoms (i.e., change score) indicates better outcome.
Hamilton Depression Rating Scale (HRSD-24) | immediately after the intervention
  The 24-item version of the Hamilton Depression Rating Scale is an established clinician-
Hamilton Depression Rating Scale (HRSD-24) | Follow-up (6 months after the intervention)
  The 24-item version of the Hamilton Depression Rating Scale is an established clinician-

SECONDARY OUTCOMES:
Patient Health Questionnaire 9 (PHQ-9) | Total Time Frame is 7 months. Outcome is assessed at three points: baseline; post-intervention and Follow-up (6 months after the intervention)]
  9-item scale developed to assess depressive symptoms and to evaluate the symptoms of depression.
Beck-Depressions-Inventar II (BDI-II) | Total Time Frame is 7 months. Outcome is assessed at three points: baseline; post-intervention and Follow-up (6 months after the intervention)]
  Change in self-assessed depression as measured by the Beck Depression Inventory (BDI) total score from baseline to post-assessment (8 weeks) and baseline to follow-up (5 months). The BDI is a 21-item self-report measure of depression symptoms. Total scores range from 0-63 with higher scores indicating more severe levels of depression.
Mini Mental State Examination (MMSE) | Total Time Frame is 7 months. Outcome is assessed at three points: baseline; post-intervention and Follow-up (6 months after the intervention)]
  Developed by Folstein et al, 1975 to assess cognitive deficits.
Dysfunctional Attitudes Scale Form 18B (DAS-18B) | Total Time Frame is 7 months. Outcome is assessed at three points: baseline; post-intervention and Follow-up (6 months after the intervention)]
  Change in dysfunctional attitudes as measured by change in the Dysfunctional Attitudes Scale Form 18B (DAS-18B) total score and subscale scores from baseline to post-assessment (8 weeks) and baseline to follow-up (5 months). Each item is endorsed on a 7-point scale (Range: 0-7) such that a total score of 126 is possible with higher scores indicating dysfunctional beliefs which are held more strongly. The total score is comprised of two subscales (perfectionism (Range 0-56); need for social approval (Range 0-21)), which are summed along with 7 other items to calculate the total scale score.
Metacognitions Questionnaire (MCQ-30) | Total Time Frame is 7 months. Outcome is assessed at three points: baseline; post-intervention and Follow-up (6 months after the intervention)]
  Change in metacognitive beliefs as measured by change in the Metacognitions Questionnaire (MCQ-30) total score and subscale scores from baseline to post-assessment (8 weeks) and baseline to follow-up (5 months). The 30-item scale has a range of 30-120. The scale is comprised of five subscales (range for each = 6-24): (1) Positive Beliefs (PB) about worry (6 items); (2) Negative Beliefs (NB) about thoughts concerning uncontrollability and danger (6 items), and (3) beliefs about the need to control thoughts (Need for Control [NFC],6 items); (4) Cognitive Confidence (6 items) and Cognitive Self-Consciousness (6 items). Higher scores indicate more strongly held metacognitive beliefs.
Rosenberg Self-Esteem Scale | Total Time Frame is 7 months. Outcome is assessed at three points: baseline; post-intervention and Follow-up (6 months after the intervention)]
  Change in self-esteem as measured by change in the Rosenberg Self-Esteem scale total score from baseline to post-assessment (8 weeks) and baseline to follow-up (5 months). The scale is comprised of 10 items and scores range from 10-40 with higher scores indicating higher self-esteem.
Ruminative Responses Scale | Total Time Frame is 7 months. Outcome is assessed at three points: baseline; post-intervention and Follow-up (6 months after the intervention)]
  Change in rumination as measured by the Ruminative Responses Scale total score from baseline to post-assessment (8 weeks) and baseline to follow-up (5 months). The scale is comprised of 10 items and scores range from 10-40 with higher scores indicating higher self-esteem.
Attitudes to Ageing Questionnaire (AAQ) | Total Time Frame is 7 months. Outcome is assessed at three points: baseline; post-intervention and Follow-up (6 months after the intervention)]
  The attitudes to ageing questionnaire (AAQ) [12] was developed to provide a standard way of measuring attitudes to ageing from the perspective of older people.
ICF Core Set for Depression | Total Time Frame is 7 months. Outcome is assessed at three points: baseline; post-intervention and Follow-up (6 months after the intervention)]
  was developed through the WHO International Classification of Functioning, Disability and Health (Cieza et al., 2004), and criteria are being developed to make the assessment more objective, through the modified e-Delphi technique.
World Health Organization Quality of Life-BREF - Item 1 | Total Time Frame is 7 months. Outcome is assessed at three points: baseline; post-intervention and Follow-up (6 months after the intervention)]
  Change in global quality of life as measured by change on item 1 on the World Health Organization Quality of Life-BREF from baseline to post-assessment (8 weeks) and baseline to follow-up (5 months). Responses on the item range from 1 (very bad quality of life) to 5 (very good quality of life).

CONTACTS AND LOCATIONS:
Locations (1):
- Lara Manuela Guedes de Pinho, Evora, Portugal

REFERENCES:
- [Derived] de Pinho LG, Silva C, Fonseca C, Morgado B, Lopes M, Moritz S, Jelinek L, Schneider BC. A randomized controlled trial to evaluate the efficacy of metacognitive training for older adults with depression (MCT-Silver) in Portugal: study protocol. Front Psychol. 2023 Oct 31;14:1167860. doi: 10.3389/fpsyg.2023.1167860. eCollection 2023. PMID 38022953